CLINICAL TRIAL: NCT07010484
Title: Using Novel Imaging to Rethink Diagnostic and Treatment Strategies for Polymyalgia Rheumatica
Acronym: REMAP PMR
Status: Recruiting | Type: Observational
Sponsor: Kresten Krarup Keller (Other)
Collaborators: Randers Regional Hospital (Other); Central Jutland Regional Hospital (Other); Gødstrup Hospital (Other); Svendborg Hospital (Other); Odense University Hospital (Other); Regionshospitalet Horsens (Other)
Responsible Party: Sponsor-Investigator, Kresten Krarup Keller, Associate professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: 1-10-72-69-25; NNF24OC0094827 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Polymyalgia Rheumatica (PMR)
Keywords: polymyalgia rheumatica; imaging; diagnosis; PET/CT; PET/MRI
MeSH Terms: conditions — Polymyalgia Rheumatica; Disease | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with and suspected of polymyalgia rheumatica: The study evaluate a new method to diagnose PMR with PET/CT using magnetic resonance imaging (MRI) for informing the interpretation of PET in 111 patients suspected of polymyalgia rheumatica (PMR) at baseline and after 8 weeks prednisolone treatment.
  In addition, a treatment initiation strategy guided by clinical diagnosis combined with PET will be evaluated in 100 patients with newly diagnosed PMR (estimated 64 from the 111 patients with suspected PMR, and additionally 38 diagnosed with PMR of which approximately 34 will have PMR without concurrent giant cell arteritis). Patients with a clinical diagnosis of PMR and a negative PET will not be started in routine treatment, but receive intramuscular glucocorticoids, which can be followed by oral prednisolone 15 mg tapered during a maximum of 3 month after diagnosis at discretion of the investigator.
  Interventions: Diagnostic Test: PET/MRI; Diagnostic Test: PET/CT with 18-FDG

INTERVENTIONS:
Diagnostic Test: PET/MRI — PET/MRI at baseline and week 8
Diagnostic Test: PET/CT with 18-FDG — PET/CT in patients not receiving PET/MRI

SUMMARY:
Polymyalgia rheumatica (PMR) is the most common chronic inflammatory rheumatic disease among the elderly and is characterized by proximal extremity pain and fatigue. Treatment with prednisolone carries several significant adverse effects, and it is therefore essential to avoid unnecessary treatment. However, clinical diagnosis and even imaging such as positron emission tomography and computed tomography (PET/CT) has low diagnostic accuracy, which decrease after start of prednisolone. The purpose is to evaluate a new method to diagnose PMR with PET/CT using magnetic resonance imaging (MRI) for informing the interpretation of PET in 111 patients suspected of PMR at baseline and after 8 weeks prednisolone treatment. In addition, a treatment initiation strategy guided by clinical diagnosis combined with PET will be evaluated in 100 patients with newly diagnosed PMR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suspected of PMR seen at the Department of Rheumatology/internal medicine in Aarhus, Silkeborg, Horsens, Gødstrup, Randers, and Svendborg.
2. Age above 50.
3. Proximal extremity pain.

Exclusion Criteria:

1. Oral, intravenous, intra-articular or intramuscular glucocorticoids within the last 2 months.
2. Previous prednisolone treatment for GCA/PMR.
3. Unable to give consent.
4. Proximal extremity pain duration for more than one year.
5. Symptoms of GCA (headache, scalp tenderness, jaw or tongue claudication, vision disturbances attributable to GCA, limb claudication).
6. Active malignant cancers within the last 5 years (except basal cell carcinoma).
7. Other known inflammatory rheumatic diseases (e.g. rheumatoid arthritis, polymyositis, spondyloarthritis, psoriatic arthritis, gout).
8. Uncontrolled diseases (e.g. severe active asthma, cardiac disease with NYHA class IV)
9. For MRI: Implants contraindicating MRI and BMI>150 kg.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected of and diagnosed with polymyalgia rheumatica are included.
Sampling Method: Probability Sample
Enrollment: 149 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Clinical diagnosis of PMR after 1 year and a positive baseline [18F]FDG-PET scan, with MRI findings used to support interpretation of the PET evaluation. | Baseline
  sensitivity and specificity of [18F]FDG-PET/CT using PET combined with MRI to inform the interpretation of the PET evaluation, using the clinical diagnosis at 1 year as reference standard.
A clinical diagnosis of PMR at baseline and a negative PET not requiring glucocorticoids for more than 3 months during the first year. | Baseline to 1 year
  proportion of patients with a positive clinical diagnosis and a negative PET not requiring glucocorticoids for more than 3 months during the first year.

SECONDARY OUTCOMES:
Clinical diagnosis of PMR after 1 year and a positive [18F]FDG-PET/MRI at baseline. | Baseline
  Sensitivity and specificity of [18F]FDG-PET/MRI at baseline for diagnosing PMR, using the clinical diagnosis at 1 year as reference standard.
Clinical diagnosis of PMR after 1 year and a positive MRI at baseline. | Baseline
  Sensitivity and specificity of MRI at baseline for diagnosing PMR, using the clinical diagnosis at 1 year as reference standard.
Circular, focal, and/or cylindrical [18F]FDG-uptake patterns associated to synovitis, bursitis, and tendinitis/tenosynovitis in the shoulders and hips on MRI or ultrasound. | Baseline
  Investigate if circular, focal and cylindrical [18F]FDG-uptake patterns correspond to synovitis, bursitis and tendinitis using MRI and ultrasound for confirmation.
Clinical diagnosis of PMR after 1 year and synovitis, bursitis, and tendinitis/tenosynovits in the shoulders and hips. | Baseline
  Prevalence of synovitis, tendinitis/tenosynovitis and bursitis in PMR and differential diagnoses.
Clinical diagnosis of PMR after 1 year and extra-capsular PMR diagnosed using [18F]FDG-PET/MRI. | Baseline
  Proportion of patients with capsular and extra-capsular PMR.
Extra-capsular PMR and remission after 2 or 4 weeks. | Baseline to 4 weeks
  Time to remission in patients with extra-capsular involvement compared to PMR patients with capsular involvement.
Extra-capsular PMR with relapse and remaining in prednisolone treatment within the first year, first 3 years, and first 5 years. | Baseline to 5 years
  Proportion of patients with capsular and extra-capsular PMR who experience relapse and remain in prednisolone treatment within the first year, first 3 years, and first 5 years.
Clinical diagnosis of PMR after 1 year and a positive [18F]FDG-PET/CT after 8 weeks of prednisolone treatment, with MRI findings used to support PET interpretation. | 8 weeks
  Sensitivity and specificity of [18F]FDG-PET after 8 weeks of prednisolone treatment using PET combined with MRI to inform the interpretation of PET scans for diagnosing PMR, using the clinical diagnosis at 1 year as reference standard.
Clinical diagnosis of PMR after 1 year and a positive [18F]FDG-PET/MRI after 8 weeks of prednisolone treatment. | 8 weeks
  Sensitivity and specificity of [18F]FDG-PET/MRI after 8 weeks of prednisolone treatment for diagnosing PMR, using the clinical diagnosis at 1 year as reference standard.
Clinical diagnosis of PMR after 1 year and a positive MRI after 8 weeks of prednisolone treatment. | 8 weeks
  Sensitivity and specificity of MRI after 8 weeks of prednisolone treatment for diagnosing PMR, using the clinical diagnosis at 1 year as reference standard.
Specific baseline clinical information and baseline, 8 weeks, or changes after 8 weeks of prednisolone treatment on [18F]FDG-PET/MRI findings, and the prediction of relapse and prednisolone-free remission after 1 year, 3 years, and 5 years. | Baseline to 5 years
  Investigate whether clinical information or [18F]FDG-PET/MRI findings at baseline, 8 weeks, or changes after 8 weeks of prednisolone treatment can predict relapse and prednisolone-free remission after 1 year, 3 years, and 5 years.
Specific baseline clinical information and baseline, 8 weeks, or changes after 8 weeks of prednisolone treatment on MRI findings, and the prediction of relapse and prednisolone-free remission after 1 year, 3 years, and 5 years. | Baseline to 5 years
  Investigate whether clinical information or MRI findings at baseline, 8 weeks, or changes after 8 weeks of prednisolone treatment can predict relapse and prednisolone-free remission after 1 year, 3 years, and 5 years.
Specific baseline clinical information and baseline, 8 weeks, or changes after 8 weeks of prednisolone treatment on ultrasonography findings, and the prediction of relapse and prednisolone-free remission after 1 year, 3 years, and 5 years. | Baseline to 5 years
  Investigate whether clinical information and ultrasonography findings at baseline, 8 weeks, or changes after 8 weeks of prednisolone treatment can predict relapse and prednisolone-free remission after 1 year, 3 years, and 5 years.
Baseline characteristics for patients with a positive PET scan and a clinical diagnosis of PMR at baseline. | Baseline
  Compare baseline characteristics between patients with a positive PET scan and a clinical diagnosis of PMR and those with a negative PET scan and a clinical diagnosis of PMR.
Baseline MRI findings for patients with a positive PET scan and a clinical diagnosis of PMR at baseline. | Baseline
  Compare MRI findings between patients with a positive PET scan and a clinical diagnosis of PMR and those with a negative PET scan and a clinical diagnosis of PMR.
Baseline characteristics for patients with a clinical diagnosis of PMR at baseline and a negative PET scan not receiving glucocorticoids for more than 3 months during the first year. | Baseline to 1 year
  Investigate if baseline characteristics can predict which patients with a clinical PMR diagnosis will have a negative PET and require glucocorticoids for no longer than 3 months during the first year.
Clinical diagnosis of PMR after 1 year and symptomatic or asymptomatic (subclinical) GCA at diagnosis, week 8, year 1, year 3, and year 5 in patients diagnosed with PMR. | Baseline to 5 years
  Prevalence of symptomatic and asymptomatic (subclinical) GCA at diagnosis, week 8, year 1, year 3 and year 5 in patients diagnosed with PMR.
Clinical diagnosis of PMR after 1 year and positive ultrasound findings around the shoulders and hips at baseline, week 8, year 1, year 3, and year 5. | Baseline to 5 years
  Changes in ultrasound findings around the shoulders and hips during 1 year, 3 years and 5 years.
Physical activity evaluated with step count using the physical activity tracking application over the course of one year in patients with PMR. | Baseline to 1 year
  Changes in physical activity during the first year after diagnosis.
Decreased physical activity during doctor-diagnosed relapses of PMR. | Baseline to 1 year
  Investigate if relapses of PMR can be detected with physical activity tracking.
Fulfilling the criteria for fibromyalgia at baseline and after 1, 3, and 5 years. | Baseline to 5 years
  Proportion of PMR patients fulfilling the criteria for fibromyalgia after 1 year, 3 years and 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Kresten K Keller, MD, PhD, Principal Investigator — Department of Rheumatology, Aarhus University Hospital
Locations (7):
- Denmark (7):
  - Aarhus University Hospital, Aarhus
  - Gødstrup Hospital, Gødstrup
  - Horsens Regional Hospital, Horsens
  - Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Central Jutland Regional Hospital, Silkeborg
  - Svendborg Hospital, Svendborg

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in the publications
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication, and 2 years.
Access Criteria: By resonably request.